CLINICAL TRIAL: NCT07258784
Title: RNA Sequencing of Discarded Tracheal Stenosis Tissue to Characterize Cellular and Molecular Pathogenesis
Status: Recruiting | Type: Observational
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Chenchen Zhang, Assistant professor, University of Maryland, Baltimore
Other Study IDs: HP-00114191
Record Dates: First submitted 2025-11-20; First posted 2025-12-02 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-09

CONDITIONS: Tracheal Stenosis; Subglottic Stenosis
MeSH Terms: conditions — Tracheal Stenosis | interventions — Biopsy; Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Biopsied or resected stenotic tissue from patients with benign tracheal stenosis
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients with benign tracheal stenosis undergoing either endoscopic or surgical treatment
  Interventions: Procedure: Biopsy or surgery

INTERVENTIONS:
Procedure: Biopsy or surgery — The tissue will be obtained from biopsy or surgical resection. All the "intervention" will be performed for clinical needs. The tissue used in the study will be considered as discarded tissue

SUMMARY:
Benign tracheal stenosis is a rare but potentially life-threatening condition, typically resulting from fibroinflammatory scarring. It can be secondary to iatrogenic etiologies such as intubation or tracheostomy , as well as autoimmune diseases and being idiopathic. Patients typically undergoes endoscopic or surgical interventions to open up the airways. This project will analyze resected or biopsied tissue from patients with benign tracheal stenosis to define disease-specific RNA expression profiles.

ELIGIBILITY:
Inclusion Criteria:

* Patients with benign tracheal stenosis

Exclusion Criteria:

* Malignancy. active infection

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with benign tracheal stenosis, including idiopathic, iatrogenic, autoimmune.
Sampling Method: Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2025-09-11 (Actual); Primary Completion 2026-09-10 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
RNA profile | 1 year
  The diseased mucosa will show a increased fibrosis and inflammation profile compared with that from normal mucosa

CONTACTS AND LOCATIONS:
Locations (1):
- University of Maryland, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided